CLINICAL TRIAL: NCT06098222
Title: The Effect of Slow Breathing Exercise Applied to Patients After Primary Percutaneous Coronary Intervention on Pulse, Blood Pressure and Quality of Life
Brief Title: The Effect of Slow Breathing Exercise Applied to Patients on Pulse, Blood Pressure and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Melike Çelik, Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TUBITAKprojectnumbered223S237; 223S237 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2023-10-05; First posted 2023-10-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Slow Breathing; Acute Myocardial Infarction
Keywords: Blood Pressure; Pulse; Percutaneous Coronary Intervention; Quality of Life; Slow Breathing Exercise
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow breathing exercise training (Experimental): Slow breathing exercise training will be given to patients in the experimental group. After discharge, patients will be asked to do slow breathing exercises twice a day for 10 minutes every day for eight weeks. Daily and/or weekly online, weekday, weekend, daytime, evening, video phone calls will be made with patients who are discharged at the end of the training to practice the slow breathing exercise every day according to the patients' demand. It will be provided that breathing exercises will be performed together with a video call in the form of a conference call. Patients will be asked to take measurements a total of two days a week, one day on weekdays and one day on weekends, in the morning, after a light breakfast, at least five minutes of rest and breathing exercises. Pulse and blood pressure measurements at home on weekdays will be asked to be measured Decouply from breathing exercise, and on weekends before and after breathing exercise.
  Interventions: Behavioral: Slow breathing exercise training
- Control group (No Intervention): In the control group, patients will be shown and told self-blood pressure and pulse measurement at home at discharge. A reminder text message will be sent to the mobile phones of patients for blood pressure and pulse measurement at home. The control group will also be asked to perform their own blood pressure and pulse monitoring at home and record a Self-Monitoring Form (for the Control group).During home follow-up, patients will be sent reminder text messages to their mobile phones two days a week. According to the request of patients, daily and/or weekly online, weekdays, weekends, daytime, evening, phone calls will be made to measure pulse and blood pressure values two days a week.

INTERVENTIONS:
Behavioral: Slow breathing exercise training — Slow breathing exercise training will be given by the researcher in a single one-hour session in the meeting room of the unit 24 hours after the PCI and/or the next day. After a 20-minute silent rest in the training, patients will be asked to breathe slowly through the nostrils for 4 seconds and slowly exhale through the mouth for 6 seconds to reach 6-8 breaths/min. The patient will rest for 5 seconds after every 6 slow breaths. During the training period, a stopwatch will be used by observing the patient's chest and abdominal movements in order to determine whether the patients have reached the required respiratory rate.
  Arms: Slow breathing exercise training

SUMMARY:
This study was designed as a randomized controlled experimental type in order to determine the effect of slow breathing exercise applied after the procedure on heart rate, blood pressure and quality of life in patients who underwent Primary Percutaneous Coronary Intervention (PCI) I after the diagnosis of ST Elevation Myocardial Infarction (STEMI).

Patients who underwent primary PCI due to STEMI in a Training and Research Hospital in Istanbul will constitute the study population. A sample will be formed with a total of 80 patients, 40 experimental and 40 control groups, selected by computer assisted simple randomization method among volunteer patients who underwent primary PCI and met the inclusion criteria.

In this study, slow breathing exercise training will be given to the experimental group by the coordinator. In their home followmup after discharge, they will be asked to do slow breathing exercises for 10 minutes twice a day for eight weeks.

Data will be collected using the "Patient Information Form", "MacNew Heart Disease Health Related Quality of Life Scale", "VAS Breath Therapy Satisfaction Evaluation Form", "Self-Monitoring Form" and "Patient Follow up Form". Patients will be seen again during the outpatient clinic examination in the fourth and eighth weeks and the effectiveness of slow breathing exercises will be evaluated with data collection forms.

DETAILED DESCRIPTION:
Cardiovascular Diseases (CVD) is still the leading cause of death in the world and in our country, despite significant advances in its diagnosis and treatment. Acute Coronary Syndromes (ACS), which are among the CVD's, occur with the deterioration of the integrity of the atherosclerotic plaque in the coronary vessels. The deadliest form of ACS is ST Elevation Myocardial Infarction (STEMI).

Primary Percutaneous Coronary Intervention (PCI) is recommended primarily in the treatment of acute myocardial infarction. In these patients, changes in vital signs resulting from diagnosis and treatment and a permanent effect on quality of life can be observed.

Slow breathing exercise is a behavioral technique in which a low breathing rate is applied. Breathing exercises reduce heart rate, blood pressure, reduce anxiety and pain while shown to improve symptoms and improve quality of life in patients with chronic obstructive pulmonary disease and asthma. This technique provides conscious deep and slow breathing and effective breathing, as well as improving conscious control over relaxation and increasing awareness.

This study was designed as a randomized controlled experimental type in order to determine the effect of slow breathing exercise applied after the procedure on heart rate, blood pressure and quality of life in patients who underwent PCI after the diagnosis of STEMI. Study data will be collected between 23 October 2023- 30 April 2024 Patients who underwent primary PCI due to STEMI in a Training and Research Hospital in Istanbul will constitute the study population. A sample will be formed with a total of 80 patients, 40 experimental and 40 control groups, selected by computer assisted simple randomization method among volunteer patients who underwent primary PCI and met the inclusion criteria.

In the study, slow breathing exercise training will be given to the experimental group by the coordinator. In their home followmup after discharge, they will be asked to do slow breathing exercises for 10 minutes twice a day for eight weeks. It will be ensured that video calls and breathing exercises are performed together in the form of conference calls.. "Slow Breathing Exercise Training Booklet" and "Slow Breathing Exercise Short Film Video" will be used in the trainings. A calibrated portable digital upper arm sphygmomanometer will be used for heart rate and blood pressure measurement. Groups will be asked to record their own pulse and blood pressure measurements at home.

Data will be collected using the "Patient Information Form", "Mac New Heart Disease Health Related Quality of Life Scale", "VAS Breath Therapy Satisfaction Evaluation Form", "Self-Monitoring Form" and "Patient Follow up Form". Patients will be seen again during the outpatient clinic examination in the fourth and eighth weeks and the effectiveness of slow breathing exercises will be evaluated with data collection forms.

SPSS (IBM Corp., Armonk, NY, USA) program will be used in the analysis of the findings. Before analysis, the normality of the data will be evaluated with the Shapiro-Wilk test. Comparisons between the two groups will be made with descriptive statistics (frequency, percentage, etc.) in the analysis, as well as the Independent Sample t-test (in data with normal distribution) and Mann-Whitney U test (in data that does not show normal distribution) in quantitative data. In comparisons of more than two groups, One-Way Analysis of Variance (One-way ANOVA) or its non-parametric equivalent Kruskal-Wallis test will be used. Paired Samples t-Test or its non-parametric equivalent Wilcoxon test will be used to test the difference in quantitative repeated measurements. Qualitative comparisons between groups will be made with the Chi-Square test. Results, significance in the 95% confidence interval will be evaluated under p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Young adult patients between the ages of 18-65,
* Patients who have not received fibrinolytic therapy before or simultaneously with Percutaneous Coronary Intervention (PCI) procedure,
* Patients who have passed 24 hours after the PCI procedure,
* Patients with a pulse > 60/min (whether or not beta blockers are used after PCI),
* Patients without rhythm problems,
* Patients with hypertension (systolic blood pressure 140-179 mmHg, diastolic blood pressure 90-109 mmHg), (whether or not they use antihypertensive and beta blocker drugs),
* Patients without a diagnosis of mental or psychiatric disease,
* Patients who have the materials to watch the breathing exercise video,
* Patients who can receive reminder messages and make video calls (with devices such as a smartphone, computer, tablet, etc.),
* Patients with a portable blood pressure monitor suitable for pulse and blood pressure measurement during home monitoring (the necessary equipment will be provided within the scope of the TUBITAK project),
* Patients without hearing or visual impairment,
* Patients who can read and write
* Patients who can communicate,
* Patients without language problems,
* Patients who volunteer and indicate this verbally and in writing

Exclusion Criteria:

* Patients with elective/appointed appointments for whom PCI is planned in advance,
* Patients whose PCI procedure failed,
* Patients who underwent only thrombus aspiration and balloon angioplasty during the PCI procedure,
* Patients who have previously undergone PCI and at least one year has not passed since,
* Patients who do not comply with planned interventions,
* Patients who do not volunteer to participate in the study,
* Patients with physical limitations and respiratory distress who cannot do breathing exercises,
* Patients with rhythm problems,
* Patients with diseases that can increase heart rate (anemia, hyperthyroidism, hyperthermia, infection),
* Patients who are morbidly obese (Body Mass Index > 40 kg/m2),
* Patients with hearing impairment,
* Patients with mental disabilities or perception problems,
* Patients who have previously received breathing therapy training will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Slow breathing exercise changes the pulse rate | 2 months
  The pulse rate in the experimental group that applied slow breathing exercises after Percutaneous Coronary Intervention is expected to be statistically significantly (p<0.05) lower than the control group.
  A calibrated portable digital upper arm blood pressure monitor purchased within the scope of the TUBITAK project will be delivered to the patient to measure pulse values.
  Volunteers will be asked to take measurements twice a week, one weekday and one weekend, in the morning, after a very light breakfast or 2 to 4 hours after a meal, and after at least five minutes of rest and breathing exercise.
  The experimental group's heart rate will be measured at home on weekdays, independently of the breathing exercise, and on the weekends, before and after the breathing exercise.
  Patients will be given a patient follow up form to record data.
Slow breathing exercise changes systolic blood pressure | 2 months
  Systolic blood pressure in the experimental group that applied slow breathing exercises after Percutaneous Coronary Intervention is expected to be statistically significantly lower (p<0.05) than the control group.
  A calibrated portable digital upper arm blood pressure monitor purchased within the scope of the TUBITAK project will be delivered to the patient to measure blood pressure values.
  Volunteers will be asked to take measurements two days a week, one weekday and one weekend, in the morning, after a very light breakfast or 2 to 4 hours after a meal, and after at least five minutes of rest and breathing exercise.
  The experimental group's blood pressure measurements will be measured at home during the weekdays, independently of the breathing exercise, and on the weekends, before and after the breathing exercise.
  Patients will be given a patient follow up form to record data.
Slow breathing exercise changes diastolic blood pressure | 2 months
  Diastolic blood pressure in the experimental group that applied slow breathing exercises after Percutaneous Coronary Intervention is expected to be statistically significantly lower (p<0.05) than the control group.
  A calibrated portable digital upper arm blood pressure monitor purchased within the scope of the TUBITAK project will be delivered to the patient to measure blood pressure values.
  Volunteers will be asked to take measurements two days a week, one weekday and one weekend, in the morning, after a very light breakfast or 2 to 4 hours after a meal, and after at least five minutes of rest and breathing exercise.
  The experimental group's blood pressure measurements will be measured at home during the weekdays, independently of the breathing exercise, and on the weekends, before and after the breathing exercise.
  Patients will be given a patient follow up form to record data.
Mac New Heart Disease Health Related Quality of Life Scale | 2 months
  Mac New Heart Disease Health Related Quality of Life Questionnaire is a scale developed by Oldridge et al. in 1991 to determine the quality of life of patients after Myocardial Infarction. This scale is designed to evaluate how physical, emotional, social functions and daily activities are affected by Coronary Artery Disease over a two week period.
  This scale consists of three subscales and 27 items: physical limitation scale (n=13), emotional function scale (n=14) and social function scale (n=13).
  Scores range from 1 to 7 on average. A low score indicates worse quality of life, a high score indicates better quality of life. Some of the items contain more than one sub-dimension. Subscale scores are calculated by averaging the answers to questions in each subscale, and considering possible scores ranging from 1 to 7, higher scores indicate a better quality of life.
  Cronbach Alpha Value is > 0.93. Written permission was obtained for the use of the scale.

SECONDARY OUTCOMES:
Satisfaction of Breathing Exercise | 2 months
  Visual Analog Scale will be used to evaluate patients' satisfaction with breathing therapy. A score of 'one' on the scale indicates that they are dissatisfied with the applied breathing therapy, a score of 'five' indicates that satisfaction is moderate, a score of '10' indicates that satisfaction is very high, and it will be indicated that satisfaction increases as the score increases. Patients will be asked to rate the level of satisfaction with breathing therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Melike CELIK, Lecturer, Principal Investigator — Marmara University; Selda CELIK, Assoc.Prof., Study Director — University of Health science; MELİKE CELİK, Lecturer, Study Chair — 905321562205
Locations (1):
- Istanbul Provincial Directorate of Health Koşuyolu High Specialization Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD sharing will be decided after the data collection has been started. It is planned to share the study protocol.

REFERENCES:
- [Derived] Celik M, Celik S. Effects of Slow Breathing Exercises on Heart Rate, Blood Pressure, and Quality of Life in Patients Undergoing Primary Percutaneous Coronary Intervention: Randomized Controlled Trial. Appl Psychophysiol Biofeedback. 2026 Feb 2. doi: 10.1007/s10484-026-09767-9. Online ahead of print. PMID 41627721